CLINICAL TRIAL: NCT00617682
Title: Maternal Immunization To Prevent Infant Otitis Media
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: George Curlin, Medical Officer, DMID, NIAID, NIH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01DC005974-03 (NIH)
Record Dates: First submitted 2008-02-14; First posted 2008-02-18 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Otitis Media
Keywords: Maternal immunization; Pneumococcal conjugate vaccine; Otitis media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Group 1 (experimental)
  Interventions: Biological: PNCRM9
- Group 2 (Placebo Comparator): Group 2 (placebo comparator)
  Interventions: Biological: Placebo comparator

INTERVENTIONS:
Biological: PNCRM9 — 0.5 mL IM at 30-35 wks gestation
  Arms: Group 1
Biological: Placebo comparator — Sucrose cake (NaCl and sucrose) in aluminum phosphate adjuvant diluent at 0.5 mg per 0.5 mL dose IM at 30-35 wks gestation
  Arms: Group 2

SUMMARY:
The main objective of this study is to evaluate whether immunization with 9-valent pneumococcal conjugate vaccine (PNCRM9) during the third trimester of pregnancy interferes with active antibody production in offspring immunized with PNCRM7 (Prevnar) in the first six months of life.

DETAILED DESCRIPTION:
There were 24.5 million physician visits for otitis media (OM) in 1990 with estimated treatment and indirect costs of $5 billion. Because of its major public health impact and the troubling increase in antibiotic resistant organisms, vaccine strategies to prevent OM are being tested. We previously proposed an efficacy study to determine if immunization with pneumococcal vaccine during pregnancy protects offspring against early infant OM, which is an important predictor for recurrent and chronic OM. Recent data from an efficacy trial in California demonstrated that infants immunized with 7-valent pneumococcal conjugate vaccine (PNCRM7) at 2, 4, 6 and 12 - 15 months were protected against invasive pneumococcal disease after 7 months of age. Since licensure of this vaccine, questions have been raised about whether maternal immunization with a pneumococcal vaccine during pregnancy suppresses active antibody production in offspring who are immunized with 7-valent pneumococcal conjugate vaccine (PNCRM7). The main objective of this study is to investigate that question. We will also evaluate vaccine safety, immunogenicity, and fetal antibody transfer among women who receive 9-valent pneumococcal conjugate vaccine (PNCRM9) at 30 - 35 weeks of pregnancy, determine persistence of maternal and infant antibody 13 months after birth, evaluate opsonic activity of maternal and infant antibody, and determine the relationship between breast milk and serum antibody in lactating women.

ELIGIBILITY:
Inclusion Criteria:

Maternal inclusion criteria:

* Pregnant, at least 18 yrs of age and healthy based on medical history.
* Plans to continue HealthPartners insurance coverage until infant is 13 mos old; mother and child will receive care in staff model clinic participating in the study, and obstetric care will be provided by a HP obstetrician/CNM with delivery at affiliated hospital.
* Plans to reside in Twin Cities metro area until infant is 13 mos old.
* Has a residence phone and a back-up phone contact.
* Provides informed consent.

Infant inclusion criteria:

* Infants born to enrolled women.

Exclusion Criteria:

Maternal exclusion criteria:

* Known hypersensitivity to any of the vaccine components or to latex.
* Prior vaccination with any S. pneumoniae vaccine.
* Recent (w/in 2 mos) vaccination with diphtheria or tetanus-diphtheria toxoid vaccines. Administration of influenza, or any other vaccine, or RhoGAM in the 2 wks prior to administration of the study product.
* Known history of life-threatening pneumococcal infection.
* Known impairment of immunologic function or history of immunodeficiency.
* Previous child with a major congenital anomaly or fetal malformation.
* Known to be carrying more than one fetus.
* Any medical condition or history that, in the opinion of the investigator, may interfere with the evaluation of the study objectives.
* History of preterm birth or fetal death.
* Known history of chronic hypertension, severe pre-eclampsia in a previous pregnancy, current pre-eclampsia or any type of diabetes mellitus.
* Known anatomical defects of the cervix or uterus.
* Known history of teratogenic drug use or illegal substance abuse during current pregnancy, not including tobacco or alcohol use.
* Women who have tested positive (based on medical record information) for HIV or hepatitis B infection.
* Any contraindication specified in the vaccine manufacturer's CIB.
* History of febrile illness (temp 100.0 degrees F or over) during the 72 hrs prior to vaccine administration.
* History of significant mental illness (e.g. schizophrenia, psychoses, major depression).

Infant exclusion criteria:

* Hypersensitivity to any component of the vaccine, including diphtheria toxoid.
* Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection.
* Latex sensitivity.
* Known impaired immune responsiveness, whether due to the use of immunosuppressive therapy (including irradiation, corticosteroids, antimetabolites, alkylating agents, and cytotoxic agents), a genetic defect, HIV infection, or other causes that may reduce antibody response to active immunization.
* Vaccination may be delayed because of a current or recent febrile illness depending largely on the severity of the symptoms and their etiology. Although a severe or even a moderate febrile illness is sufficient reason to postpone vaccinations, minor illnesses, such as a mild upper respiratory infection with or without low-grade fever, are not generally contraindications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2000-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Determine if offspring of women immunized with PNCRM9 or control during the third trimester have equivalent anticapsular polysaccharide (PS) IgG antibody responses to PNCRM7 measured 1 mo after the 3rd injection given at 6 mos of age. | In infants at 7 months of age; In women at 1-7 days post-immunization

SECONDARY OUTCOMES:
Determine if offspring of these women have equivalent antibody responses to PNCRM7 at 13 mos. Sera are analyzed for anti-PS IgG, opsonic activity, IgG1 & IgG2 subclasses (14,6B,19F,23F), & antibodies against Hib-PRP & diphtheria toxoid. | In infants at 13 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Ferrieri, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - HealthPartners Research Foundation, Bloomington, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Background] Le CT, Grambsch PM, Giebink GS. Quality control and the identification of vaccine responders using ELISA-derived antibody data. Stat Med. 2003 Sep 30;22(18):2935-42. doi: 10.1002/sim.1530. PMID 12953289
- [Background] Daly KA, Toth JA, Giebink GS. Pneumococcal conjugate vaccines as maternal and infant immunogens: challenges of maternal recruitment. Vaccine. 2003 Jul 28;21(24):3473-8. doi: 10.1016/s0264-410x(03)00354-2. PMID 12850363
- [Derived] Daly KA, Scott Giebink G, Lindgren BR, Knox J, Haggerty BJ, Nordin J, Goetz S, Ferrieri P. Maternal immunization with pneumococcal 9-valent conjugate vaccine and early infant otitis media. Vaccine. 2014 Dec 5;32(51):6948-6955. doi: 10.1016/j.vaccine.2014.10.060. Epub 2014 Oct 30. PMID 25444821